CLINICAL TRIAL: NCT02038998
Title: Unicentric, Phase II, Randomized Study Comparing Periodic Acceleration Versus Static Position in Cerebrovascular Stroke Patients
Brief Title: Randomized Study Comparing Periodic Acceleration Versus Static Position in Cerebrovascular Stroke Patients
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Lack of available patients
Sponsor: Fundacion Rioja Salud (Other)
Collaborators: Hospital San Pedro de Logroño (Other)
Responsible Party: Principal Investigator, Alfredo Martinez, Group Leader, Fundacion Rioja Salud
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CIBIR002
Record Dates: First submitted 2013-12-30; First posted 2014-01-17 (Estimated); Last update posted 2023-02-15 (Actual); Status verified 2021-10

CONDITIONS: Cerebrovascular Stroke
Keywords: stroke; periodic acceleration; endothelium release; ischemic penumbra; shear stress; adrenomedullin
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Static group (Sham Comparator): Control group. They will receive the standard care provided by the protocols of the ictus unit. They will lay on the Exer-Rest® TL device but the acceleration will NOT be connected.
  Interventions: Device: Exer-Rest® TL
- Single pGz intervention (Experimental): In addition to the standard care established in the ictus unit, these patients will receive a single exposure to pGz on the Exer-Rest® TL, for 3 hours, during the first day of their stay in the hospital.
  Interventions: Device: Exer-Rest® TL
- Multiple pGz interventions (Experimental): In addition to the standard care, these patients will be exposed to 45 minutes of pGz, on the Exer-Rest® TL, every day during their first week in the Hospital.
  Interventions: Device: Exer-Rest® TL

INTERVENTIONS:
Device: Exer-Rest® TL — Exer-Rest® TL is a therapeutic motorized platform that allows the application of pGz forces to a patient. The typical application would provide an acceleration of 0.4 Gz.

SUMMARY:
Stroke is one of the leading causes of death and disability worldwide. More than 85% of strokes are due to blood vessel occlusion resulting in partial destruction of the brain parenchyma. Current protocols try to re-establish blood circulation as soon as possible through chemical and/or mechanical interventions but new strategies are needed.

Periodic acceleration (pGz) is a non-invasive method consisting in the application of a rocking movement to the patient that ultimately will induce the release of beneficial chemicals from the vascular endothelium (the cells lining the inside of the blood vessels). Application of pGz in an animal model of stroke resulted in a dramatic reduction of associated brain damage.

This trial will investigate whether stroke patients exposed to pGz experiment significantly higher recovery than patients that remained static during their treatment.

DETAILED DESCRIPTION:
Periodic acceleration (pGz) is a non-invasive method consisting in the application of a rocking movement to the patient that ultimately will induce the release of beneficial chemicals from the vascular endothelium (the cells lining the inside of the blood vessels). Application of pGz in an animal model of stroke resulted in a dramatic reduction of associated brain damage.

This trial will investigate whether stroke patients exposed to pGz experiment significantly higher recovery than patients that remained static during their treatment.

ELIGIBILITY:
Inclusion Criteria:

* A signed informed consent form must be obtained prior to recruitment
* Patients with symptoms of acute ischemic stroke
* Less than 12 hours from initiation of the stroke
* Age: 18 years or older
* Capable of following the protocol

Exclusion Criteria:

* Pregnant or lactating women, and women that do not follow a contraceptive plan and may become pregnant
* Less than 18 years of age
* More than 12 hours from the initiation of the stroke or when the initiation time is unknown.
* Hemorrhagic stroke
* Candidates to receive thrombolytic treatment
* Spine traumatism or other conditions that may be aggravated by pGz
* Patients that cannot be properly followed because of phycological, social, familiar, or geographical reasons.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2015-01 (Actual); Primary Completion 2022-05 (Actual); Study Completion 2022-06 (Actual)

PRIMARY OUTCOMES:
NIHSS and Rankin scales | 0hr, 2hr, 24hr, 48hr, 7ds, 90ds
  The NIHSS and Rankin scales will be applied to the patients at the indicated times

SECONDARY OUTCOMES:
Infarct volume | 7 days
  Infarct volume will be measured by nuclear magnetic resonance 7 days after stroke

OTHER OUTCOMES:
Blood markers | 0, 1, 3, 5, and 7ds
  Neuroprotective substances that can be released by pGz (nitric oxide, tissue plasminogen activator, adrenomedullin, prostaglandins, etc) will be measured in the blood of patients to investigate the efficacy of the treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Francisco Julian-Villaverde, MD, Principal Investigator — Hospital San Pedro de Logroño; Alfredo Martinez, PhD, Study Director — Fundacion Rioja Salud
Locations (1):
- Hospital San Pedro, Logroño, La Rioja, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Martinez-Murillo R, Serrano J, Fernandez AP, Martinez A. Whole-body periodic acceleration reduces brain damage in a focal ischemia model. Neuroscience. 2009 Feb 18;158(4):1390-6. doi: 10.1016/j.neuroscience.2008.12.005. Epub 2008 Dec 14. PMID 19135137